CLINICAL TRIAL: NCT05667519
Title: Prevention of Pacemaker Lead Induced Tricuspid regurgitAtion by Transesophageal eCho guidEd Implantation (PLACE)
Acronym: PLACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Daniel Braun, MD, Senior attending physician department of cardiology, principal investigator, LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PLACE
Record Dates: First submitted 2022-12-02; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Tricuspid Regurgitation; Pacemaker Complication
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transesophageal echocardiography + fluoroscopy guided lead implantation (Experimental): TEE will be done in addition to fluoroscopy to guide lead implantation.
  Interventions: Procedure: Additional guidance of lead implantation by transesophageal echocardiography
- Fluoroscopy guided lead implantation (No Intervention): Fluoroscopy only will be used to guide lead implantation.

INTERVENTIONS:
Procedure: Additional guidance of lead implantation by transesophageal echocardiography — Transesophageal echocardiography guidance of lead implantation targeting a stable lead position in a tricuspid valve commissure (preferentially postero-septal) and an apical ventricular lead position
  Arms: Transesophageal echocardiography + fluoroscopy guided lead implantation

SUMMARY:
This is the first randomized controlled trial comparing transesophageal echocardiography + fluoroscopy guided lead implantation vs. standard lead implantation guided by fluoroscopy only. Patients are randomized 1:1 in the two groups and followed up for up to 3 years.

DETAILED DESCRIPTION:
Lead-induced tricuspid regurgitation is a frequent complication after pacemaker- and ICD-implantation that is associated with increased mortality and hospitalizations for heart failure. Transesophageal echocardiography has shown to be a safe and feasible way to guide right ventricular lead placement and was associated with less worsening of tricuspid regurgitation than standard lead implantation in a small study with a retrospective control group. This is the first randomized controlled trial comparing transesophageal echocardiography + fluoroscopy guided lead implantation vs. standard lead implantation guided by fluoroscopy only. Patients are randomized 1:1 in the two groups and followed up for up to 3 years. Echocardiographic grading of the primary endpoint will be performed by a blinded echocardiographer according to current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* indication for right ventricular lead implantation according to current guidelines

Exclusion Criteria:

* preexisting tricuspid regurgitation ≥ grade 2
* other severe heart valve disease
* history of tricuspid valve treatment
* preexisting right ventricular lead
* chronic dialysis
* contraindication for transesophageal echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Worsening of tricuspid regurgitation by at least one grade | Mean follow up of 2 years
  Worsening of tricuspid regurgitation by at least one grade on transthoracic echocardiography according to current guidelines

SECONDARY OUTCOMES:
Death and cardiovascular death | Mean follow up of 2 years
  All cause death and cardiovascular death
Heart failure hospitalizations | Mean follow up of 2 years
  Unplanned hospitalizations for heart failure
Duration of procedure and radiation | Mean follow up of 2 years
  Standard parameters affecting quality of device implantation
Right ventricular function and geometry as assessed by transthoracic echocardiography | Mean follow up of 2 years
  Right ventricular function (TAPSE, fractional area change, 3D volumetry) and geometry as assessed by transthoracic echocardiography
Sensing, Pacing and RV-stimulation of the right ventricular lead | Mean follow up of 2 years
  Sensing, Pacing and RV-stimulation of the right ventricular lead in the pacemaker readout
Change in functional capacity as assessed NYHA classification | Mean follow up of 2 years
  New York Heart Association (NYHA) Functional Classification
Change in quality of life as assessed by MLHFQ | Mean follow up of 2 years
  Minnesota Living with Heart Failure Questionnaire

OTHER OUTCOMES:
Safety Endpoint | During hospital stay (up to day 7)
  Freedom from esophageal injury, pericardial effusion and pneumothorax requiring intervention as well as lead infection/-displacement requiring lead revision

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Braun, MD, Principal Investigator — LMU Klinikum
Locations (1):
- LMU Klinikum, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No